CLINICAL TRIAL: NCT02251691
Title: The Influence of Once-daily Versus Twice-daily Immunosuppressive Regimen on Drug Compliance in Patients After Renal Transplantation
Brief Title: Influence of Once-daily Versus Twice-daily Immunosuppressant on Renal Transplant
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Astellas Pharma Taiwan, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201401105MIPA
Record Dates: First submitted 2014-06-15; First posted 2014-09-29 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Adherence to Medication Regime
Keywords: Compliance
MeSH Terms: conditions — Medication Adherence; Patient Compliance | interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Advagraf (Experimental): Take Advagraf once daily
  Interventions: Drug: Advagraf
- Prograf (Active Comparator): Take tacrolimus twice daily
  Interventions: Drug: Prograf

INTERVENTIONS:
Drug: Advagraf — Compare the drug compliance between once daily or twice daily regimen
  Other Names: Advagraf once daily
  Arms: Advagraf
Drug: Prograf — Compare the drug compliance between once daily or twice daily regimen
  Other Names: Prograf twice daily
  Arms: Prograf

SUMMARY:
The main objective of this study was to compare the drug compliance in patients after renal transplantation under once or twice-daily tacrolimus-based immunosuppressive regimen.

The rationale for this study is to access the influence of once-daily prolonged-release tacrolimus versus standard twice-daily tacrolimus on drug compliance in renal transplantation recipients base on the assumption that once-daily dosing regimen may help to improve drug compliance.

DETAILED DESCRIPTION:
This study will be a prospective, two-arm randomized and open-label, phase IV study to compare the drug compliance in patients under prolonged-release once-daily tacrolimus versus standard twice-daily tacrolimus based regimen after de novo renal transplantation.

The investigators will evaluate the drug compliance of the patients under once or twice-daily tacrolimus-based regimen using the medication scale BAAIS® (basal assessment of adherence with immunosuppressive medication scale)

ELIGIBILITY:
Male and female adult patients who are to receive renal transplantation may enter the study. The intention is to enroll 90 patients who have fulfilled inclusion/exclusion criteria into the study. Sixty patients will receive prolonged-release once-daily tacrolimus based therapy; the other thirty patients will receive standard twice-daily tacrolimus based therapy.

Inclusion criteria

* Male or female patients at 20-65 years of age undergoing renal transplantation
* Patients who have been informed of the potential risks and side effects of the study
* Female patients of childbearing potential must agree to maintain effective birth control during the study.
* Patients have been fully informed and have given written informed consent to participate in the study

Exclusion criteria

* Donor age greater than 65 years
* Patients receiving a perfectly matched kidney (6 matches HLA-A, B, DR)
* Patients who are recipients of multiple solid organ transplants
* Patients undergoing second or subsequent transplantation
* Patients with pre-transplant PRA > 20%
* Patients with ABO incompatibility or positive lymphocytotoxicity
* Patients with severe, active infection
* Patients who have an abnormal liver profile such as ALT, AST, alkaline phosphatase or total bilirubin >3 times the upper normal limit
* Patient who are HIV-positive or hepatitis C (PCR+ only) B surface antigen positive
* Patients who have been treated with an investigational drug or therapy within one month prior to entry or who will be so treated within 6 months of transplantation
* Patients with a history of malignancy within the last five years except excised squamous or basal cell carcinoma
* Patients with a history of alcohol or drug abuse or signs of alcohol-induced organ damage, mental dysfunction or other factors limiting their ability to comply fully with the study requirements.
* Patients who require on-going dosing with a systemic immunosuppressive drugs prior to transplantation.
* Pregnant woman or breast-feeding mother during the period of this study.
* Patients who are allergy to tacrolimus, macrolide antibiotics, steroid or mycophenolate mofetil.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-05-09 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
basal assessment of adherence with immunosuppressive medication scale | 12 months
  We will evaluate the drug compliance of the patients under once or twice-daily tacrolimus-based regimen using the medication scale BAAIS® (basal assessment of adherence with immunosuppressive medication scale)

SECONDARY OUTCOMES:
serum creatinine level | 12 months
  We will evaluate the serum creatinine level of the patients enrolled in this study.
graft survival | 12 months
  We will evaluate the graft survival of the patients enrolled in this study.
patient survival | 12 months
  We will evaluate the patient survival of the patients enrolled in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Yuan Lee, Principal Investigator — hospital medical school affiliations
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829